CLINICAL TRIAL: NCT03631797
Title: L'Etude préopératoire de la Microcirculation Pour la prédiction Des Complications après Une Chirurgie Cardiaque Sous Circulation Extracorporelle.
Brief Title: Preoperative Evaluation of Microcirculation for Prediction of Complications After Cardiac Surgery
Acronym: MONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A2341-54
Record Dates: First submitted 2018-07-30; First posted 2018-08-15 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2021-06

CONDITIONS: Extracorporeal Circulation; Complications
Keywords: Thoracic Surgery; Microcirculation; Endothelium, vascular; Microvascular reactivity; Laser Speckle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microvascular reactivity evaluation (Experimental): Patients referred for a preoperative arterial palmar arches assessment before cardiac valvular or coronary surgery.
  Intervention is measurement of microvascular reactivity with a laser speckle contrast imaging before surgery.
  Interventions: Procedure: Microvascular reactivity evaluation

INTERVENTIONS:
Procedure: Microvascular reactivity evaluation — Microcirculation will be evaluated for each patient before surgery with a laser speckle contrast imaging (LSCI) placed on the forearm. Tests will be performed for evaluation of endothelium reactivity: Iontophoresis.

SUMMARY:
Cardiac surgery is responsible for many complications. Microcirculation is involved in many of them. The objective of this study is to prospectively investigate the prognostic value of preoperative microcirculatory assessment in patients scheduled for cardiac surgery with CPB for the occurrence of postoperative complications.

Microvascular dysfunction is suspected of being involved in postoperative psycho-cognitive decline. The influence of microcirculation on the evolution of psycho-cognitive assessment is also analyzed in this study.

DETAILED DESCRIPTION:
Eligible patients are included during the preoperative assessment. Written consent is signed after complete explanation of the protocol.

Patient characteristics as treatments, medical history, and EuroSCORE II are registered. Moreover, intraoperative data is collected. Psycho-cognitive and functional evaluation is made preoperatively.

Microcirculation is evaluated for each patient before surgery. Complications are registered at the end of hospital stay. Psycho-cognitive and functional evaluation is repeated by call 30 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Valvular ou coronary elective cardiac surgery under cardiopulmonary bypass
* Fair skin phototype
* Ability to understand the study goal, no dementia.
* Affiliation to the French National Healthcare System
* Voluntary patients who have signed an informed consent

Exclusion Criteria:

* Emergency surgery
* Multiple procedures, combined surgery (valvular and coronary)
* Single aortic surgery
* Patient already included in the study (second surgery)
* Patients protected by decision of law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Postoperative complication | 30 postoperative days
  Composite criteria and include microcirculation postoperative complications:
  * Late surgical re-intervention (greater than 12 hours) for evacuation of pericardial effusion (seeps),
  * Surgical wound disunion or surgical site infection,
  * Organ failure: SOFA score greater than 2 at 48h,
  * Postoperative confusion: assessed using the Confusion Assessment Method (CAM) or the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU),
  * Acute renal failure ≥ stage 2 according to the KDIGO classification,
  * Acute lung injury defined as PaO2 <55mmHg in ambient air, PaO2 / FiO2 ratio <250 or Pulse Oxygen Saturation (SpO2) <90% and need for oxygen therapy,
  * Atrial fibrillation (excluding patients with permanent Atrial Fibrillation preoperatively),
  * Hepatocellular injury (Cytolysis > 10N, Prothrombin rate and Factor V decreased < 60%).

SECONDARY OUTCOMES:
Evolution of degree of disability | Inclusion and 30 days after surgery
  Change of modified Rankin scale
Functional evolution | Inclusion and 30 days after surgery
  Change of ADL score
Mood evolution | Inclusion and 30 days after surgery
  Change of brief Geriatric Depression Scale
Cognitive evolution | Inclusion and 30 days after surgery
  Change of Mc Nair test

CONTACTS AND LOCATIONS:
Overall Officials: Samir HENNI, MD PhD, Principal Investigator — UH Angers
Locations (1):
- UH Angers, Angers, France

REFERENCES:
- [Derived] Abrard S, Streichenberger A, Riou J, Hersant J, Rineau E, Jacquet-Lagreze M, Fouquet O, Henni S, Rimmele T. Preoperative endothelial dysfunction for the prediction of acute kidney injury after cardiac surgery using cardiopulmonary bypass: a pilot study based on a second analysis of the MONS study. Perioper Med (Lond). 2024 Feb 29;13(1):12. doi: 10.1186/s13741-024-00364-0. PMID 38424616
- [Derived] Abrard S, Fouquet O, Riou J, Rineau E, Abraham P, Sargentini C, Bigou Y, Baufreton C, Lasocki S, Henni S. Preoperative endothelial dysfunction in cutaneous microcirculation is associated with postoperative organ injury after cardiac surgery using extracorporeal circulation: a prospective cohort study. Ann Intensive Care. 2021 Jan 7;11(1):4. doi: 10.1186/s13613-020-00789-y. PMID 33411095